CLINICAL TRIAL: NCT01842789
Title: Post Market Evaluation of the Acessa System With Targeting Animation Guidance (TAG)
Brief Title: Post Market Evaluation of Acessa With TAG
Acronym: TAG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results to date adequately demonstrated user preference and recovery time. Time to target (Part II) was not studied. .
Sponsor: Acessa Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CP-00-0021
Record Dates: First submitted 2013-04-17; First posted 2013-04-30 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2016-02

CONDITIONS: Uterine Fibroids
Keywords: Acessa; Fibroids; Halt; Targeting Animation; Image Overlay; Radiofrequency Ablation; RFA
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acessa Procedure w/o TAG (Other): Acessa Procedure without the use of Targeting Animation Guidance
  Interventions: Device: Acessa Procedure
- Acessa Procedure with TAG (Other): Acessa Procedure with Targeting Animation Guidance
  Interventions: Device: Acessa Procedure

INTERVENTIONS:
Device: Acessa Procedure — Acessa Procedure
  Other Names: TAG; Halt Procedure; GFA

SUMMARY:
The purpose of this study is to test both user preference and speed of targeting with the use of the Acessa System with Targeting Animation Guidance (TAG).

DETAILED DESCRIPTION:
The intent of the TAG system is to assist the gynecologist in getting the tip of the Acessa Handpiece to the fibroid by creating an animated image overlay of the movements and placement.

The study will be conducted in two parts:

Part 1: User Preference Testing - users will be presented with various statements pertaining to the features of the system and asked to indicate their degree of agreement.

Part 2: Time to target - will be measure by fibroid.

ELIGIBILITY:
Inclusion Criteria: Women who:

* Are planning to undergo the Acessa procedure
* Are willing and able to comply with all procedures
* Are capable of providing informed consent

Exclusion Criteria: Women who:

* In the medical judgement of the investigator should not participate in this study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Galen, MD, Principal Investigator — Donald I Galen Consulting
Locations (1):
- Donald I Galen Consulting, San Ramon, California, United States

REFERENCES:
- [Background] Hayhurst C, Byrne P, Eldridge PR, Mallucci CL. Application of electromagnetic technology to neuronavigation: a revolution in image-guided neurosurgery. J Neurosurg. 2009 Dec;111(6):1179-84. doi: 10.3171/2008.12.JNS08628. PMID 19326991
- [Background] Fried MP, Parikh SR, Sadoughi B. Image-guidance for endoscopic sinus surgery. Laryngoscope. 2008 Jul;118(7):1287-92. doi: 10.1097/MLG.0b013e31816bce76. PMID 18391767
- [Background] Krucker J, Xu S, Glossop N, Viswanathan A, Borgert J, Schulz H, Wood BJ. Electromagnetic tracking for thermal ablation and biopsy guidance: clinical evaluation of spatial accuracy. J Vasc Interv Radiol. 2007 Sep;18(9):1141-50. doi: 10.1016/j.jvir.2007.06.014. PMID 17804777
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Lee BB. Laparoscopic ultrasound-guided radiofrequency volumetric thermal ablation of symptomatic uterine leiomyomas: feasibility study using the Halt 2000 Ablation System. J Minim Invasive Gynecol. 2011 May-Jun;18(3):364-71. doi: 10.1016/j.jmig.2011.02.006. PMID 21545960
- [Background] Bergamini V, Ghezzi F, Cromi A, Bellini G, Zanconato G, Scarperi S, Franchi M. Laparoscopic radiofrequency thermal ablation: a new approach to symptomatic uterine myomas. Am J Obstet Gynecol. 2005 Mar;192(3):768-73. doi: 10.1016/j.ajog.2004.10.591. PMID 15746670
- [Background] Milic A, Asch MR, Hawrylyshyn PA, Allen LM, Colgan TJ, Kachura JR, Hayeems EB. Laparoscopic ultrasound-guided radiofrequency ablation of uterine fibroids. Cardiovasc Intervent Radiol. 2006 Jul-Aug;29(4):694-8. doi: 10.1007/s00270-005-0045-9. PMID 16502165
- [Background] Robles R, Aguirre VA, Argueta AI, Guerrero MR. Laparoscopic radiofrequency volumetric thermal ablation of uterine myomas with 12 months of follow-up. Int J Gynaecol Obstet. 2013 Jan;120(1):65-9. doi: 10.1016/j.ijgo.2012.07.023. Epub 2012 Oct 14. PMID 23073229
- [Background] Chudnoff SG, Levine DJ, Galen DI, et al. Prospective 12-month follow up of quality-of-life improvement following 135 consecutive cases laparoscopic and ultrasound-guided radiofrequency ablation of fibroids. J Minim Invasive Gynecol. 2012;19(Suppl):S45.
- [Background] Lee BB. Radiofrequency ablation of uterine fibroids; a new minimally invasive hysterectomy alternative. Obstet Gynecol. 2002;99(Suppl):S9.
- [Background] Chudnoff SG, Berman JM, Levine DJ, Harris M, Guido RS, Banks E. Outpatient procedure for the treatment and relief of symptomatic uterine myomas. Obstet Gynecol. 2013 May;121(5):1075-1082. doi: 10.1097/AOG.0b013e31828b7962. PMID 23635746
- [Background] Macer JA. For uterine-sparing fibroid treatment, consider laparoscopic ultrasound-guided radiofrequency ablation. obmanagement.com Vol 25 No. 11 November 2013
- [Result] Galen DI. Electromagnetic image guidance in gynecology: prospective study of a new laparoscopic imaging and targeting technique for the treatment of symptomatic uterine fibroids. Biomed Eng Online. 2015 Oct 15;14:90. doi: 10.1186/s12938-015-0086-5. PMID 26471917

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acessa Procedure w/o TAG | Acessa Procedure With TAG
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acessa Procedure w/o TAG | Acessa Procedure With TAG | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Full Range); unit: Years] | 41.8 [28.5 to 49.6] | 43.9 [31.2 to 52.9] | 42.7 [28.5 to 52.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician Feedback Regarding TAG System Use During Surgery.
Description: Physician preference testing is assessed by the completion of a questionnaire using a 5 point rating system ranging from "strongly agree" (a rating of 5) to "strongly disagree" (a rating of 1) regarding the use of the TAG system. The questions included are in regards to ease of targeting, ease of visualizing the target, the addition of specific features that enhance user interface and the overall set-up.
Time Frame: Physicians have up to 1 hour after the procedure to fill out the questionnaire
Population: All subjects in whom TAG was used as an accessory system. This outcome measure was specific to this arm of the study only. Physicians provided feedback regarding use of the accessory system but did not provide feedback regarding the standard system without guidance. Physicians rated the system on a scale of 1 Strongly disagree to 5 Strongly agree.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acessa Procedure With TAG
Number analyzed (Participants) | 8
units on a scale
  Transducer and handpiece dynamic animation was | 5.0 (0)
  The use of TAG enabled the ability to reach the fi | 5.0 (0)
  Knowing the handpiece trajectory helped to tar | 5.0 (0)
  The transducer and handpiece dynamic animation hel | 4.7 (0.46)
  The use of TAG provided confidence when targeting | 4.9 (0.35)

2. Primary Outcome: Number of Minutes From Visualizing the Target to Reaching the Target
Description: To measure difference in time to target with and without the use of TAG. This is a time and motion study, with time measured at each stage of the procedure. The most important subject variable to consider was number of fibroids targeted, which influenced overall procedure time.
Time Frame: Intraoperative
Population: All participants undergoing treatment with Acessa (with or without targeting animation guidance).
Measure: Mean (Full Range); unit: Minutes per fibroid treated
Arm/Group | Acessa Procedure w/o TAG | Acessa Procedure With TAG
Number analyzed (Participants) | 10 | 8
Minutes per fibroid treated | 29.9 [8.9 to 65.0] | 25.2 [15.1 to 45.0]

3. Secondary Outcome: Recovery Time
Description: Patients to be followed for 1 to 2 months post-treatment to evaluate recovery.
Time Frame: 1 to 2 months
Population: All subjects followed for 1 to 2 months post treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Acessa Procedure w/o TAG | Acessa Procedure With TAG
Number analyzed (Participants) | 10 | 6
days | 8.5 [2 to 45] | 6 [4 to 21]

ADVERSE EVENTS:
Time Frame: 30 days post operative follow up
Arm/Group | Acessa Procedure w/o TAG | Acessa Procedure With TAG
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/8
Other Adverse Events (participants affected / at risk) | 0/10 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acessa Procedure w/o TAG (N=10) | Acessa Procedure With TAG (N=8)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — obstruction of the lower bowel approximately one month after the Acessa procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acessa Procedure w/o TAG (N=10) | Acessa Procedure With TAG (N=8)
Poor wound healing (Skin and subcutaneous tissue disorders) | 0 | 1 — For one subject, the Acessa procedure incision was found to be not healing properly approximately 10 days after the procedure. The severity of this complication was considered moderate, treated with medications, and resolved appropriately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No